CLINICAL TRIAL: NCT05115864
Title: The Role of Self-assessment Combined with Home-based Wearable Device Over Supervised Pelvic Floor Muscle Training for Stress or Mixed Urinary Incontinence in Postpartum Women: a Multi-center Randomized Controlled Trial
Brief Title: Comparison Between Home-based Wearable Device and Supervised PFMT on SUI/MUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFMT-PUMCH
Record Dates: First submitted 2021-11-02; First posted 2021-11-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-03

CONDITIONS: Stress Urinary Incontinence
Keywords: pelvic floor muscle training; stress urinary incontinence; wearable device
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PFMT with device (intervention) group (Experimental): The patients in PFMT with device (intervention) group followed the practice program three months. During three months, the intervention group is commanded to complete the PFMT program with the vaginal device and assess the grade of type I and II pelvic floor muscle fiber strength once three weeks.
  Interventions: Device: PFMT with device
- PFMT alone （control） group (No Intervention): The patients in PFMT alone (control) group are commanded to follow the same practice program three months without using the device.

INTERVENTIONS:
Device: PFMT with device — The wearable PFMT device (XFT-0010CK) is made by two parts. One part is the screen device which is able to show the real-time vaginal resting pressure and voluntary contraction pressure in units of mmHg. The other part is a vaginal air-filled probe. The two parts are combined with a thin air tube. The whole device is connected to a smartphone app by Bluetooth to record the progress of PFMT. There are two modes of the device, one is assessment mode, when it comes to the assessment mode that the device is able to assess the grade of type I and II pelvic floor muscle fiber strength by the patients themselves, the other mode is practice mode by displaying real-time visual pressure value according to the completeness of the PFMT program.
  Arms: PFMT with device (intervention) group

SUMMARY:
Objective The study is designed to compare the benefit of self-assessment of a home-based wearable device assisted pelvic floor muscle training (PFMT) to standard supervised PMFT program for women with SUI/MUI (stress urinary incontinence/mixed urinary incontinence).

Background National and international clinical practice guidelines recommend supervised pelvic floor muscle training of at least 3 months' duration as a first-line treatment to women (including the elderly and post-natal) with stress or mixed urinary incontinence (Level of evidence A). However, it remains unknown that which component could bring extra benefit when assisted with surprised PFMT.

Patients selection and study design The study protocol was approved by the Peking union medical college hospital ethics committee (JS-3192D, 26/10/2021). Women who had their 6-week to 3-month postpartum clinical visits in the member hospitals between Dec 01, 2021 and May 01, 2022 were invited to participate in the study. The women who reported SUI/MUI symptoms within 3 months postpartum were recruited. The exclusion criteria were 1）urgency urinary incontinence alone; 2）a prolapse greater than stage II on examination (>1cm below the hymen on straining); 3）third and fourth degree perineal tear; 4）suffering diastasis recti abdominis and chronic pelvic pain as the primary problem need treatment; 5）a history of stress urinary incontinence(SUI) before pregnancy; 6）had previous pelvic surgery; 7）malignant pelvic cancer; 8）Genurological infection; 9）had received formal instruction on PFMT in the past 5 years; 10）unsuitable to participate because of significant diseases; 11）others:were unable to contract pelvic floor muscles on digital examination when requested;Inability to use the device in vagina. Once each participate was recruited, they were arranged randomly to either an intervention group or a control group (1:1). The intervention group used a wireless wearable vaginal device to record the pressure and practice time and the grade of type I and II pelvic floor muscle fiber strength were assessed by the device once three weeks. The control group accepted the supervised PFMT. Both groups followed the same program three months. During three months, the investigators phoned both groups once three weeks to guide their training. Both groups were assessed by questionnaire and PFM measurements at baseline(pre-test), 3-month, 6-month and 12-month. The primary outcome is ICIQ-UI SF; The secondary outcomes include POP-SS; POP-Q; Oxford Classification; Pelvic floor muscle surface electromyography; I-QOL; PISQ-12; BPMSES.

The hypothesis is that the wearable device with self-assessment function providing PFMT is superior to the supervised PFMT program alone for the treatment of both SUI and MUI of postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks<After delivery<3 mo postpartum
* Clinically diagnosed stress or mixed urinary incontinence as the primary problem
* Women aged 18 years or older

Exclusion Criteria:

* Urgency urinary incontinence alone
* A prolapse greater than stage II on examination (>1cm below the hymen on straining)
* Third and fourth degree perineal tear;
* Suffering diastasis recti abdominis and chronic pelvic pain as the primary problem need treatment
* A history of stress urinary incontinence (SUI) before pregnancy
* Had previous pelvic surgery
* Malignant pelvic cancer
* Genitourinary system infection
* Had received formal instruction on PFMT in the past 5 years
* Unsuitable to participate because of significant diseases
* Others: were unable to contract pelvic floor muscles on digital examination when requested; Inability to use the device in vagina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire [ICIQ-UI SF] | Baseline (pre-test)
  The ICIQ-UI SF score ranges from 0 to 21 and is the weighted sum of three items addressing urinary incontinence frequency ("how often do you leak urine?" 0=never to 5=all the time), leakage quantity ("how much urine do you usually leak?" 0=none to 6=a large amount), and interference with everyday life (0=not at all to 10=a great deal). Higher scores reflect greater severity.
Change from Baseline ICIQ-UI SF at 3 months | at 3 months
  The change on the severity of SUI
Change from Baseline ICIQ-UI SF at 6 months | at 6 months
  The change on the severity of SUI
Change from Baseline ICIQ-UI SF at 12 months | at 12 months
  The change on the severity of SUI

SECONDARY OUTCOMES:
Quality-of-life outcomes: Incontinence Quality of Life Instrument [I-QOL] | at baseline(pre-test), 3-month, 6-month and 12-month
  The instrument has 3 subscales: (1) avoidance and limiting behavior, (2) psychosocial impacts, and (3) social embarrassment. All items are evaluated using a 5-point Likert-type scale. The 22 items in the I-QOL were summed and transformed to a 0 to 100 scale for greater interpretability, with the higher scores representing better quality of life.
Pelvic floor-related outcomes: Pelvic Organ Prolapse Symptom Score [POP-SS] | at baseline(pre-test), 3-month, 6-month and 12-month
  POP-SS contains seven items relating to frequency of prolapse symptoms. Each item is scored from 0 (never) to 4 (all the time), with a possible total score ranging from 0 to 28. Higher scores reflect greater severity.
Sex function outcome: the short-form Prolapse Incontinence Sexual Questionnaire [PISQ-12] | at baseline(pre-test), 3-month, 6-month and 12-month
  Ranging from 0 to 48, with higher scores indicating greater sexual dysfunction
Self-efficacy outcomes:Chinese version of the broome pelvic muscle self-efficacy scale: reliability and validity[BPMSES] | at baseline(pre-test), 3-month, 6-month and 12-month
  It is a 23-item rating scale consisting of two domains: efficacy expectations and outcome expectations. In efficacy expectations domain, participants demonstrate how confident they are in performing pelvic floor muscle training. In outcome expectations domain, participants show the confidence that the training will prevent unwanted urine leakage. The score ranges are from 0 to 100. The higher the score, the greater self-efficacy perceived by the participant.
The Pelvic Organ Prolapse Quantification (POP-Q) | at baseline(pre-test), 3-month, 6-month and 12-month
  The Pelvic Organ Prolapse Quantification (POP-Q) approach was used to measure the positions of vaginal structures relative to the hymenal ring. Stage of POP was diagnosed using the reliable and valid Pelvic Organ Prolapse-Quantification examination (POP-Q) in which the maximal point of vaginal descent is measured relative to the hymen during strain with the woman in the 45-degree lithotomy position.
Oxford grading scale | at baseline(pre-test), 3-month, 6-month and 12-month
  It consists of a six-point scale ranging from 0 to 5, 0 indicating no muscle activity, 1 minor muscle flicker, 2 weak muscle activity, 3 moderate muscle contraction, 4 good muscle contraction and 5 a strong muscle contraction
PFM strength assessed by manometry | at baseline(pre-test), 3-month, 6-month and 12-month
  The outcomes included vaginal resting pressure (VRP), maximum vaginal pressure (MVP), maximum voluntary contraction pressure (MVCP), the grade of type I and II pelvic floor muscle fiber strength.
Patient adherence to treatment | During the 3-month supervised treatment
  In our study, patients' adherence to treatment will be determined as the frequency of exercises anticipated for 3 months of supervised treatment, which will be subjectively self-reported and objectively device-recorded. Patients' overall adherence will be categorized as follows: 50%≤= low adherence; 50%-75%= medium adherence; and ≥75%= high adherence.
Patient Global Impression of Improvement (PGI-I) | at 3, 6, 9, and 12 weeks during 3-month intervention
  Answers to the question "which best describes your urinary symptoms now, compared with how they were before this study" are evaluated on a seven-point scale ranging from 1 = Very much better to 7 = Very much worse. Only answers affirming a score of 1 (very much better) or 2 (much better) will be considered to indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuqi Wang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication including both primary and secondary outcomes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting 6 months after publication
URL: http://www.chictr.org.cn

REFERENCES:
- [Derived] Wang X, Qiu J, Li D, Wang Z, Yang Y, Fan G, Mao X, Wang J, Gao S, Zhu X, Xu T, Sun Z. Pressure-Mediated Biofeedback With Pelvic Floor Muscle Training for Urinary Incontinence: A Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2442925. doi: 10.1001/jamanetworkopen.2024.42925. PMID 39499517
- [Derived] Wang X, Sun Z, Xu T, Fan G. Efficacy of supervised pelvic floor muscle training with a home-based biofeedback device for urinary incontinence in postpartum women: protocol for a multicentre randomised controlled trial. BMJ Open. 2023 Apr 25;13(4):e069874. doi: 10.1136/bmjopen-2022-069874. PMID 37185188